CLINICAL TRIAL: NCT06194474
Title: Study on Biomarkers of Postoperative Delirium in Elderly Cardiac Surgery Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jining First People's Hospital (Other)
Responsible Party: Principal Investigator, Fuhui Yan, Study Director, Jining First People's Hospital
Other Study IDs: JNFPH-2023-01
Record Dates: First submitted 2023-12-16; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Delirium Group
- No Delirium Group

SUMMARY:
To evaluate the relationship between abnormal protein or metabolite expression levels in peripheral blood and postoperative delirium in elderly patients undergoing cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

1. patients between 55 and 80 years old,
2. American Society of Anesthesiologists (ASA) physical status of II-III and New York Heart Association grade of II-III.
3. The planned cardiac surgery.
4. Hospitalization duration not less than 5 days.
5. The anesthesia time will be no less than 2 hours.All patients had a normal ability to hear, read and cooperate with neuropsychological tests.

Exclusion Criteria:

1. The pre-operative Montreal Cognitive Assessment (MoCA) score was less than 25,
2. Patients with dementia, history of neurological or psychiatric disease, hospital with anxiety depression scale (HADS) over eight points,
3. Currently use sedatives or antidepressants, Patients with substance dependence on drugs or alcohol.
4. Patients with liver and kidney dysfunction, patients with a history of cardiac surgery.
5. Admitted to the ICU for more than two days within the month preceding the current surgery,
6. Unable to cooperate with researcher's investigations.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To evaluate the relationship between abnormal protein or metabolite expression levels in peripheral blood and postoperative delirium in elderly patients undergoing cardiac surgery.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2022-09-05 (Actual); Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Proteomics | 1 month
  Proteomic data will be obtained by LC-MS/MS Analysis-DIA(Data Independent Acquisition) platform

CONTACTS AND LOCATIONS:
Locations (1):
- Fuhui Yan, Jining, Shandong, China